CLINICAL TRIAL: NCT03468530
Title: Therapeutic Effects of Endoscopic Ablation of Hunner Lesions in Interstitial Cystitis/ Bladder Pain Syndrome Patients
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, Professor, Samsung Medical Center
Other Study IDs: 2017-08-005
Record Dates: First submitted 2017-12-13; First posted 2018-03-16 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Transurethral ablation — transurethral resection and/or coagulation with a bipolar loop under spinal or general anesthesia

SUMMARY:
efficacy of endoscopic ablation of Hunner lesions in patients with IC/BPS and the characteristics of HLs based on a long-term follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 18 yrs or greater
2. Patients diagnosed with BPS(Bladder Pain Syndrome)
3. Symptom persisted more than 6 months
4. Pain VAS ≥4
5. O'Leary-Sant Interstitial Cystitis questionnaire (IC-Q) scores 12 or greater with pain and nocturia domain scores > 2.
6. Pelvic Pain and Urgency/Frequency Patient Symptom Scale(PUF) >13
7. No history of cystoscopy within 2yrs.

Exclusion Criteria:

1. History of augmentation cystoplasty or previous transurethral coagulation/resection due to BPS
2. Child-bearing potential, pregnant or nursing women.
3. Mean voided volume lesser than 40ml or over than 400ml.
4. Hematuria exceeds 1+ in the urinary dipstick (dipstick) examination.
5. Urinary tract infection during run-in periods.
6. Genitourinary tuberculosis or bladder,urethral and prostate cancer
7. Recurrent urinary tract infection
8. History of hysterectomy,mid-urethral sling,pelvic organ prolapse repair,vaginal delivery or Cesarean section,prostate operation or treatment etc within 6months.
9. Neurologic disease history of cerebral infarction,multiple sclerosis or parkinsonism etc.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 442 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
change in recurrence-free survival time after ablation treatment | Every three months for one year

SECONDARY OUTCOMES:
changes in mean number of daytime frequency episodes | Every three months for one year
changes in mean number of nocturia episodes | Every three months for one year
changes in mean number of urgency episodes | Every three months for one year
Change score of O'Leary-Sant Interstitial Cystitis questionnaire (IC-Q) | Every three months for one year
Score of Global Response Assessment (GRA), Patient Global Assessment (PGA) score | every 3months for one year
Change score of Pelvic Pain and Urgency/Frequency Patient Symptom Scale(PUF) | Every three months for one year
Change score of Brief Pain Inventory-short form (BPI-sf) | Every three months for one year
Occurrence of adverse event | Every three months for one year

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No